CLINICAL TRIAL: NCT05749341
Title: A Pilot Study of Liquid Biopsy Diagnostic Techniques for Endometriosis
Brief Title: A Liquid Biopsy Diagnostic Techniques for Endometriosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wenwen Wang, associate professor, Tongji Hospital
Other Study IDs: V1
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Liquid Biopsy; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Identify endometrial cell from peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Three-Dimensional Poly(dimethylsiloxane) Scaffold — The rest blood samples from patients with and without endometriosis (No. 20 VS 20) would be collected for testing on a Microchip Embedded with Three-Dimensional Poly(dimethylsiloxane) Scaffold.

SUMMARY:
To evaluate the diagnostic efficiency of circulating endometrial cell detection method using microfluidic chip as an non-invasive method for diagnosis in endometriosis.

DETAILED DESCRIPTION:
Endometriosis is a chronic condition, characterized by the presence of functional endometrial glands and interstitium in extrauterine ectopia. Ectopic endometrial tissue responds to estradiol and other hormones similar to normal endometrium. Endometriosis is one of the most common benign gynaecological conditions, affecting up to 5 to 10 percent of women of reproductive age. In addition to severe dysmenorrhea or pelvic pain, decreased fertility is a common clinical manifestation of internal heterogeneity, with up to 40 percent of patients associated with infertility . Currently, laparoscopy is the gold standard for diagnosis. However, the actual time to diagnosis in patients with internal dysmorphia is delayed by an average of 4 to 11 years, resulting in a large number of patients with moderate to severe (stage III to IV) at diagnosis. Recently, the exploration of efficient and cost-effective non-invasive diagnostic solutions has been a hot button issue.

ELIGIBILITY:
Inclusion Criteria:

• Surgically and pathologically verified patients with or without endometriosis

Exclusion Criteria:

* suspicion of malignancy
* pregnancy
* acute infection
* Lack of ability to sign informed consent forms on their own

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Planned number of sample for each group: 20 with endometriosis and 20 without endometriosis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of cases with identified circulating endometrial cells. | within one week after blood sample collecting
  To evaluate the ability of the Three-Dimensional Poly(dimethylsiloxane) Scaffold to isolating circulating endometrial cells (CEC) in patients with and without endometriosis.
  In each group, the percentage of cases with identified circulating endometrial cells will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: WENWEN WANG, DOCTOR, Study Director — Huazhong University of Science and Technology
Locations (1):
- Wenwen Wang, Wuhan, Hubei, China